CLINICAL TRIAL: NCT02888899
Title: Percutaneous Tibial Nerve Stimulation in Combination With Biofeedback in Patients With Fecal Incontinence - A Randomized Controlled Trial
Brief Title: Tibial Nerve Stimulation in Combination With Biofeedback
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Jenny Sjödahl, PhD, RPT, University Hospital, Linkoeping
Purpose: Treatment
Other Study IDs: Dnr 2015/443-31
Record Dates: First submitted 2016-08-23; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Biofeedback, Psychology; Loperamide; Karaya Gum; ispaghula seed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment (Experimental)
  Interventions: Behavioral: Biofeedback; Drug: Loperamide; Drug: Stool bulking agent (sterculia or ispaghula husk)
- PTNS in addition to standard treatment (Experimental)
  Interventions: Behavioral: Biofeedback; Drug: Loperamide; Drug: Stool bulking agent (sterculia or ispaghula husk); Other: PTNS

INTERVENTIONS:
Behavioral: Biofeedback
Drug: Loperamide
Drug: Stool bulking agent (sterculia or ispaghula husk)
Other: PTNS
  Arms: PTNS in addition to standard treatment

SUMMARY:
Background: Fecal incontinence (FI) affects 2-13% of an adult general population. The prevalence increases with age, and after 50 years of age prevalence rates up to 26% in women have been reported. Quality of life in patients with FI is decreased considerably, in a similar extent as in patients with ulcerative colitis in relapse.

Management of FI usually involves a stepwise approach; beginning with more conservative strategies and moving on to more appropriately tailored medications, bowel-retraining, biofeedback and psychosocial support. Although a combination of these treatment alternatives often improves symptoms they are not always successfully. Neuromodulation is a relatively new treatment modality for FI that is based on recruitment of residual anorectal neuromuscular function pertinent to continence by electrical stimulation of the peripheral nerve supply. Sacral Nerve Stimulation (SNS) is one type of neuromodulation and it employs direct electrical stimulation of the sacral nerves. Recently an alternative neuromodulation technique to SNS has been developed in treating FI i.e. tibial nerve stimulation. The tibial nerve contains afferent and efferent fibers originating from the forth and the fifth lumbar nerves and the first, second and third sacral nerves. Thus, stimulation of the tibial nerve may lead to changes in anorectal neuromuscular function similar to those observed with SNS but without the need of a permanent surgically implanted device. Tibial nerve stimulation is therefore an attractive treatment alternative for FI patients since the treatment is well-tolerated and treatment results have been very promising.

Aim: The overall aim is to measure the effect of percutaneous tibial nerve stimulation (PTNS) in combination with biofeedback on symptoms in consecutive FI patients compared with biofeedback alone. The investigators also aim to study which FI patients have most profit of the addition of PTNS.

Methods: The study will take place at the Pelvic Floor Unit, department of Gastroenterology, University Hospital Linköping. Prior to the first visit to the hospital a symptom diary will be mailed to the FI patients and they are instructed to record their FI symptoms, bowel habits and gastrointestinal symptoms prospectively on a 24-hour diary during 2 weeks. Before consideration of enrolment into the study, gastroenterologists assess all the patients' medical history and perform a physical examination. Subjects will also have an endoanal ultrasonography and the investigators will measure rectal volumes, sensational thresholds and anal sphincter function.

FI patients who fulfil inclusion criteria will then be randomly assigned to either PTNS in combination with biofeedback or biofeedback alone. The treatment will be performed by physiotherapists.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age with fecal incontinence for more than 6 months
* Patients with at least one or more episodes of fecal incontinence during a period of 2 weeks as recorded by bowel function diary
* Patients from whom written consent was obtained

Exclusion Criteria:

* Previous congenital or acquired spinal injury, spinal tumour or spinal surgery
* Presence of neurological diseases or peripheral vascular disease
* Uncontrolled diabetes mellitus
* Congenital anorectal malformations
* Colorectal or gastrointestinal surgery ≤24 months
* Presence of external full-thickness rectal prolapse
* Inflammatory bowel disease
* Chronic diarrhoea
* Use of tibial nerve or sacral nerve stimulations
* Ongoing pregnancy
* Any malignant disease
* Pacemaker
* Ongoing or earlier treatment with sacral- or tibial nerve stimulation
* Chronic varicose ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Change in fecal leakage episodes with a symptom diary | Change from baseline in fecal leakage episodes at 12 weeks (post-treatment), change from baseline in fecal lekage episodes at 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Sjödahl, PhD, RPT, Principal Investigator — University Hospital in Linkoeping
Locations (1):
- Pelvic floor unit, University Hospital in Linköping, Linköping, Sweden